CLINICAL TRIAL: NCT03664752
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Vehicle-Controlled, 2 Arm, Parallel Group Study Comparing the Safety and Efficacy of IDP-120 Gel and IDP-120 Vehicle Gel in the Treatment of Acne Vulgaris
Brief Title: Study Comparing the Safety and Efficacy of IDP-120 Gel and IDP-120 Vehicle Gel in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V01-120A-302
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Results first posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: Multi-Center, Randomized, Double-Blind, Vehicle-Controlled, 2 Arm, Parallel Group Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor) As a double-blinded study, the investigators, the site staff, the sponsor, and the clinical monitors will not be aware of the treatment assigned to the individual study subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IDP-120 Gel (Experimental): IDP-120 Gel, once-daily application
  Interventions: Drug: IDP-120 Gel
- IDP-120 vehicle gel (Placebo Comparator): IDP-120 vehicle gel, once daily application
  Interventions: Drug: IDP-120 Vehicle Gel

INTERVENTIONS:
Drug: IDP-120 Gel — IDP-120 Gel, once-daily application
  Arms: IDP-120 Gel
Drug: IDP-120 Vehicle Gel — IDP-120 Vehicle Gel, once-daily application
  Arms: IDP-120 vehicle gel

SUMMARY:
study designed to assess the safety, tolerability, and efficacy of IDP-120 Gel and IDP-120 Vehicle Gel

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, vehicle-controlled, 12-week study designed to assess the safety, tolerability, and efficacy of IDP-120 Gel and IDP-120 Vehicle Gel at Weeks 2, 4, 8, and 12. To be eligible for the study subjects must be at least 9 years of age and have a clinical diagnosis of moderate to severe acne

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 9 years of age and older;
2. Written and verbal informed consent must be obtained. Subjects less than age of consent must sign an assent for the study and a parent or a legal guardian must sign the informed consent (if subject reaches age of consent during the study they should be re-consented at the next study visit);
3. Subject must have a score of 3 (moderate) or 4 (severe) on the Evaluator's Global Severity Score (EGSS) assessment at the baseline visit;
4. Subjects with facial acne inflammatory lesion (papules, pustules, and nodules) count no less than 20 but no more than 50;
5. Subjects with facial acne non-inflammatory lesion (open and closed comedones) count no less than 25 but no more than 100;
6. Subjects with two or fewer facial nodules

Exclusion Criteria:

1. Use of an investigational drug or device within 30 days of enrollment or participation in a research study concurrent with this study;
2. Any dermatological conditions on the face that could interfere with clinical evaluations such as acne conglobata, acne fulminans, secondary acne, perioral dermatitis, clinically significant rosacea, gram-negative folliculitis, dermatitis, eczema;
3. Any underlying disease(s) or some other dermatological condition of the face that requires the use of interfering topical or systemic therapy or makes evaluations and lesion count inconclusive;
4. Subjects with a facial beard or mustache that could interfere with the study assessments;
5. Subjects with more than two (2) facial nodules;
6. Evidence or history of cosmetic-related acne

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 585 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — Bausch Health Companies
Locations (20):
- United States (18):
  - Valeant Site 210, Rogers, Arkansas
  - Valeant Site 201, Manhattan Beach, California
  - Valeant Site 206, San Diego, California
  - Valeant Site 218, San Diego, California
  - Valeant Site 204, Boynton Beach, Florida
  - Valeant Site 217, Brandon, Florida
  - Valeant Site 202S, Miami, Florida
  - Valeant Site 214, Tampa, Florida
  - Valeant Site 222, Snellville, Georgia
  - Valeant Site 215, Boise, Idaho
  - Valeant Site 205, Metairie, Louisiana
  - Valeant Site 216, Clarkston, Michigan
  - Valeant Site 221, Clinton Township, Michigan
  - Valeant Site 227, Rochester, New York
  - Valeant Site 229, Raleigh, North Carolina
  - Valeant Site 230, Raleigh, North Carolina
  - Valeant Site 213, San Antonio, Texas
  - Valeant Site 223, Spokane, Washington
- Canada (2):
  - Valeant Site 219, Waterloo, Ontario
  - Valeant Site 228, Waterloo, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IDP-120 Gel | IDP-120 Vehicle Gel
Started | 293 | 292
Completed | 244 | 241
Not Completed | 49 | 51

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDP-120 Gel | IDP-120 Vehicle Gel | Total
Number analyzed (Participants) | 293 | 292 | 585
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.8 (8.35) | 20.2 (7.59) | 20.5 (7.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178 | 181 | 359
  Male | 115 | 111 | 226
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 11 | 17 | 28
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 36 | 42 | 78
  White | 229 | 215 | 444
  More than one race | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Mean Lesion Counts at Week 12
Description: For noninflammatory facial lesions, open comedones (blackheads) and closed comedones (whiteheads) were recorded as a single count. For inflammatory facial lesions, papules (solid, elevated lesion less than 5 mm) and pustules (elevated lesion containing pus less than 5 mm) were recorded as a single count, while nodular lesions (palpable subcutaneous lesion greater than 5 mm) were counted and recorded separately.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Deviation); unit: lesion counts
Arm/Group | IDP-120 Gel | IDP-120 Vehicle Gel
Number analyzed (Participants) | 293 | 292
lesion counts
  Inflammatory lesion count | -18.5 (9.50) | -13.8 (9.80)
  Non-inflammatory lesion count | -26.9 (14.71) | -16.7 (15.26)

2. Primary Outcome: Percentage of Subjects Who Had at Least a 2-grade Reduction From Baseline at Week 12 in the Evaluator's Global Severity Score (EGSS) and Had an EGSS at Week 12 That Equated to "Clear" or "Almost Clear"
Description: Evaluator's Global Severity Score (EGSS) was determined based on evaluator-blinded evaluations of the signs and symptoms of acne vulgaris. Evaluations were scored on a scale of 0-4, with 0 being clear and 4 being severe.
Time Frame: Baseline to Week 12
Measure: Number; unit: percentage of participants
Arm/Group | IDP-120 Gel | IDP-120 Vehicle Gel
Number analyzed (Participants) | 293 | 292
percentage of participants | 33.2 | 14.2

3. Secondary Outcome: Percentage Change in Mean Lesion Counts at Week 12
Description: as for outcome 1
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Deviation); unit: percentage change
Arm/Group | IDP-120 Gel | IDP-120 Vehicle Gel
Number analyzed (Participants) | 293 | 292
percentage change
  Non-inflammatory lesion count | -61.82 (34.013) | -39.01 (35.025)
  Inflammatory lesion count | -64.88 (32.929) | -49.17 (34.002)

4. Secondary Outcome: Percentage of Subjects Who Had at Least a 2-grade Reduction From Baseline at Week 12 in the Evaluator's Global Severity Score (EGSS)
Description: as for outcome 2
Time Frame: Baseline to Week 12
Measure: Number; unit: percentage of participants
Arm/Group | IDP-120 Gel | IDP-120 Vehicle Gel
Number analyzed (Participants) | 293 | 292
percentage of participants | 36.8 | 16.7

5. Secondary Outcome: Percentage Change in Mean Lesion Counts at Week 8
Description: as for outcome 1
Time Frame: Baseline to Week 8
Measure: Least Squares Mean (Standard Deviation); unit: percentage change
Arm/Group | IDP-120 Gel | IDP-120 Vehicle Gel
Number analyzed (Participants) | 293 | 292
percentage change
  Non-inflammatory lesion count | -52.41 (35.796) | -28.61 (37.772)
  Inflammatory lesion count | -55.48 (32.992) | -38.42 (34.413)

6. Secondary Outcome: Percentage Change in Mean Lesion Counts at Week 4
Description: as for outcome 1
Time Frame: Baseline to Week 4
Measure: Least Squares Mean (Standard Deviation); unit: percentage change
Arm/Group | IDP-120 Gel | IDP-120 Vehicle Gel
Number analyzed (Participants) | 293 | 292
percentage change
  Non-inflammatory lesion count | -41.15 (32.860) | -23.15 (34.548)
  Inflammatory lesion count | -45.06 (32.313) | -31.37 (33.789)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | IDP-120 Gel | IDP-120 Vehicle Gel
All-Cause Mortality (participants affected / at risk) | 0/293 | 0/292
Serious Adverse Events (participants affected / at risk) | 1/293 | 2/292
Other Adverse Events (participants affected / at risk) | 53/293 | 8/292
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IDP-120 Gel (N=293) | IDP-120 Vehicle Gel (N=292)
Abortion induced (Surgical and medical procedures) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IDP-120 Gel (N=293) | IDP-120 Vehicle Gel (N=292)
Application site pain (General disorders) | 39 | 6
Application site dryness (General disorders) | 27 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor for details.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/52/NCT03664752/Prot_SAP_000.pdf